CLINICAL TRIAL: NCT05887102
Title: Pilot Study of a Community Pharmacy-Based Program to Enhance Adherence to Adjuvant Endocrine Therapy Among Breast Cancer Survivors
Brief Title: Pilot Study of PACHA Program to Enhance Adherence to Adjuvant Endocrine Therapy Among Breast Cancer Survivors
Acronym: PACHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Quebec Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: number CIHR 420809
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast Cancer; Adjuvant Endocrine Therapy; Adherence to Treatment; Community Pharmacy; Support; Survivorship; Intervention Evaluation; Pilot Study; Randomized Controlled Trial; Feasibility Study; Mixed-Methods
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled pilot trial using mixed methods (quantitative and qualitative). A cluster consists of a pharmacy, its pharmacists and its patients with adjuvant endocrine therapy (AET) prescription who have agreed to participate. Participating pharmacies will be randomly assigned to two groups. In the first group, pharmacists will provide usual services to women (control group). In the second group, pharmacist and women will have access to the PACHA program in addition to the usual services (intervention group).
Who Masked: Outcomes Assessor
Masking Description: Pharmacists and women will not be blind to the intervention but analyses of data self-reported by the participants (questionnaires) will be conducted in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACHA program group (Experimental): Pharmacists and women in the PACHA program group will receive the PACHA program component's.
  Interventions: Behavioral: PACHA Program
- Usual care group (No Intervention): Pharmacists and women in the Usual care group will provide/receive usual care.

INTERVENTIONS:
Behavioral: PACHA Program — Pharmacists in this group will complete the 85-minutes web-based training, schedule and realize at least 2 telephone consultations with participating women in their pharmacy (in the first month and 4 months after randomization) using standardized consultation guides based on the principles of motivational interviewing and, if necessary, the evidence-based web sheets about strategies to cope with side effects and other AET-related concerns. Women in this group will have access to a web site that includes video capsules to inform women about AET, evidence-based web sheets describing strategies to cope with side effects and other AET-related concerns, testimonies of women who had breast cancer and an AET and a list of resources available for women.
  Arms: PACHA program group

SUMMARY:
The goal of this randomized controlled pilot study is to assess the feasibility, acceptability, and preliminary effects of the PACHA program designed for women having an adjuvant endocrine therapy (AET) after hormone-sensitive breast cancer. PACHA (programme en Pharmacie pour l'ACcompagnement des femmes ayant de l'Hormonothérapie Adjuvante) is a community pharmacy-based program aimed at optimizing the experience of AET and its use. The main questions it aims to answer are :

* Does the program have an effect on factors expected to influence AET adherence?
* Is the program acceptable?
* Is the implementation of the program feasible?
* What is the feasibility of procedures for carrying out a full-scale study?

Participating community pharmacies will be randomized. Pharmacists working in pharmacies assigned to the PACHA group (33 pharmacies) will receive web-based training and manuals to use during their consultations with women having an AET. Recruited women attending these pharmacies will also have access to information and resources about AET (videos, evidence-based booklet). Pharmacists practicing in pharmacies assigned to the control group (33 pharmacies) will provide usual care.

DETAILED DESCRIPTION:
This is a cluster randomized controlled pilot trial using mixed methods (quantitative and qualitative). A cluster consists of a pharmacy, its pharmacists and its patients with adjuvant endocrine therapy (AET) prescription who have agreed to participate. Participating pharmacies will be randomly assigned to two groups. In the first group, pharmacists will provide usual services to women (control group). In the second group, pharmacist and women will have access to the PACHA program in addition to the usual services (intervention group).

The PACHA program consists, for the pharmacists, of:

* A 85-minutes web-based training to prepare the pharmacists for delivery of the intervention. The program comprises three main sections led by experts: 1) a review of AET pharmacotherapy; 2) information on AET consultation based on the principles of motivational interviewing and video simulations of AET consultations according to program tools and expert feedback of these simulations, and 3) access to materials geared to participating women (web-video capsules about AET, self-management strategies for coping with specific AET side effects and list of resources). The web-based training can be completed in one or more sessions. Pharmacists who complete the program will receive continuing education credits. The PACHA pharmacists will have to complete this program in the weeks after randomization.
* Standardized consultation guide based on motivational interviewing to guide AET consultations (by phone or in person). This standardized consultation guide outlines the key steps that the pharmacist must cover during the AET consultation and follows the usual sequence of consultation in pharmacy. This consultation guide is to be used in the first month and 4 months after randomization, or more frequently according to a woman's situation.
* Evidence-based web sheets describing (non)pharmacological strategies to cope with side effects (e.g. hot flashes) and other AET-related concerns (e.g. sexuality) and to guide the consultation.

For the women, the PACHA program consists of:

* Web video capsules to inform women about AET. These video capsules cover how to and why take tamoxifen or an aromatase inhibitor, the possible side effects and strategies to cope with these side effects and, finally, medication intake and daily activities (e.g. diet). This also includes testimonies of women who had breast cancer and an AET.
* Evidence-based web sheets describing (non)pharmacological strategies to cope with side effects (e.g. hot flashes) and other AET-related concerns (e.g. sexuality) in a version adapted for the woman.
* List of web resources available for women to help cope with side effects and other AET-related concerns.

Participation in the study will take place over a period of 6 months. The study will be carried out in approximately 66 pharmacies in the Quebec province (33 will be assigned to the control group and 33 to the intervention group), which include approximately 132 women (66 in the control group and 66 in the intervention group). At the end of the follow-up, pharmacists and women in the control group can, if desired, receive certain tools offered in the intervention group.

Pharmacists and participating women will be asked to completed two questionnaires: the first before randomization and the second at the end of the follow-up 6 months later.

At the end of the study, 20-30 pharmacists and 20-30 patients will be invited to take part in a semi-directed individual interview (qualitative component) in order to gather their point of view and their experience with the care and services received in relation to AET.

The characteristics of pharmacies, pharmacists and patients in the intervention and control groups will be compared. Indicators of acceptability and feasibility will be measured (e.g. recruitment and participation and retention rates). Generalized Estimating Equation (GEE) regression models will be used to compare patterns of changes in scores of factors expected to influence AET experience and adherence in the two groups and between study entry and 6 months later. The main analyzes will be performed on a intention-to-treat basis. For the qualitative component, a thematic analysis will be carried out based on the transcriptions of the semi-structured interviews. The quantitative and qualitative results will be used to optimize the PACHA program, its implementation and to design, if the results support this, a large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

For pharmacies :

* In the province of Quebec, Canada
* At least one pharmacist agrees to take charge of the project in their pharmacy
* At least one women has initiated adjuvant endocrine therapy (AET) in the last 6 months in the pharmacy

For pharmacists :

* Practicing in a pharmacy in the province of Quebec
* Provide consent

For women :

* 18 years old or older
* Were diagnosed with a first non-metastatic, hormone-sensitive breast cancer
* Received and AET prescription for the first time in the last 6 months
* Are fluent in French
* Have internet access
* Provide consent

Exclusion Criteria:

For women :

• Live in a residential facility where AET is not self-managed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to the end of 6-month follow-up in intention to adhere to adjuvant endocrine therapy | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (4 items, score range: 1-7), higher score means higher intention to adhere
Mean change from baseline to the end of 6-month follow-up in adjuvant endocrine therapy knowledge | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (17 items, score range: 0-17), higher score means higher level of knowledge
Mean change from baseline to the end of 6-month follow-up in attitude towards adjuvant endocrine therapy | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (4 items, score range: 1-7), higher score means more positive attitude
Mean change from baseline to the end of 6-month follow-up in perceived social support | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (3 items, score range: 1-7), higher score means higher level of perceived social support
Mean change from baseline to the end of 6-month follow-up in perceived behavioural control | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (4 items, score range: 1-7), higher score means higher level of perceived behavioural control
Mean change from baseline to the end of 6-month follow-up in anticipated regret | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (6 items, score range: 1-7), higher score means higher level of anticipated regret
Mean change from baseline to the end of 6-month follow-up in coping planning | Baseline and 6-month post-randomisation
  Measured by a questionnaire developed and validated by our team (6 items, score range: 1-7), higher score means higher level of coping planning
Mean change from baseline to the end of 6-month follow-up in fear of recurrence | Baseline and 6-month post-randomisation
  Measured by the Fear of cancer recurrence inventory (FCRI) severity scale (9 items, score range: 0-36), higher score means higher level of fear of recurrence
Mean change from baseline to the end of 6-month follow-up in side effects | Baseline and 6-month post-randomisation
  Measured by the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire (19 items, score range: 0-100), higher score means higher level of side effects
Mean change from baseline to the end of 6-month follow-up in the cognitive representations of medication | Baseline and 6-month post-randomisation
  Measured by the Beliefs about Medicines Questionnaire (BMQ) (5 items for specific necessity, 5 items for specific concerns, score range: 5-25, higher score means higher level of necessity or concerns
Percentage of pharmacists who used PACHA tools in the intervention group | From Baseline to 6-month post-randomisation
  Measured by a questionnaire developed by our team and collected automatically by the study website
Percentage of women who used PACHA tools | From Baseline to 6-month post-randomisation
  Measured by a questionnaire developed by our team and collected automatically by the study website
Mean number of interventions dispensed by the pharmacists to the participating women | From Baseline to 6-month post-randomisation
  Measured by a questionnaire developed by our team and collected automatically by the study website
Percentage of eligible and enrolled pharmacists | Baseline
  Percentage
Percentage of eligible and enrolled women | Baseline
  Percentage
Percentage of pharmacies randomized | Baseline
Cluster size | Baseline
  Size

SECONDARY OUTCOMES:
Proportion of days covered by an Adjuvant Endocrine Therapy (AET) | From Baseline to 5 years post-randomisation
  Measured by a questionnaire developed by our team and analysis of AET dispensing collected via pharmacy records
Proportion of women having an AET | From Baseline to 5 years post-randomisation
  Measured by a questionnaire developed by our team and analysis of AET dispensing collected via pharmacy records
Mean change from baseline to the end of 6-month follow-up in quality of life | From Baseline to 6-month post-randomisation
  Measured by the Short-Form-12 (SF-12) questionnaire
Program Acceptability and Feasibility | At the end of 6-month follow-up (post-randomisation)
  Measured by semi-structured interviews conducted with pharmacists and participating women on the relevance, acceptability and perceived benefits of each program component (intervention group only).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dionne, B.Pharm., M.Sc., Study Director — Laval University; Michel Dorval, Ph.D., Study Director — Laval University; Line Guénette, Ph.D., Study Director — Laval University; Jason Guertin, Ph.D., Study Director — Laval University; Laurence Guillaumie, Ph.D., Study Director — Laval University; Lyne Lalonde, Ph.D., Study Director — Université de Montréal; Julie Lemieux, MD,M.Sc., Study Director — CHU de Québec-Université Laval; Benoît Masse, Ph.D., Study Director — St. Justine's Hospital; Hermann Nabi, Ph.D., Study Director — Laval University; Louise Provencher, MD, Study Director — CHU de Québec-Université Laval
Locations (1):
- Centre de recherche du CHU de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lapointe J, Guillaumie L, Dionne A, Lalonde L, Lemieux J, Dorval M, Nabi H, Lemay M, Guenette L, Guertin JR, Masse B, Lauzier S. A community pharmacy-based program to enhance adherence to adjuvant endocrine therapy among breast cancer survivors (PACHA): protocol for a pilot cluster-randomized controlled trial. Pilot Feasibility Stud. 2025 Jul 14;11(1):98. doi: 10.1186/s40814-025-01676-8. PMID 40660375